CLINICAL TRIAL: NCT03560843
Title: The Effect of Mindfulness Based Stress Reduction (MBSR) on Patients With Traumatic Brain Injury and Chronic Insomnia
Brief Title: The Effects of MBSR on Patients With TBI and Chronic Insomnia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 900001
Record Dates: First submitted 2018-03-13; First posted 2018-06-18 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Chronic Insomnia; TBI (Traumatic Brain Injury)
Keywords: MBSR, TBI, insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: MBSR is an 8 week standardized protocol that includes gentle yoga, meditation, and mindfulness practices that were originally developed by Jon Kabat-Zinn from the University of Massachusetts. A trained MBSR instructor will lead group sessions weekly for approximately 150-210 minutes to teach and demonstrate the practices. Practices include walking/standing/supine meditation, body scanning (drawing attention to various areas of the body such as the right foot or left hand), and simple hatha yoga postures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBSR treatment (Experimental): MBSR will be administered over 8 week period.
  Interventions: Behavioral: MBSR
- Control group (No Intervention): Usual care will continue for this group.

INTERVENTIONS:
Behavioral: MBSR — Mindfulness Based Stress Reduction
  Arms: MBSR treatment

SUMMARY:
To evaluate the effects of Mindfulness Based Stress Reduction (MBSR) as an adjunct to usual clinical care for treatment of stress and chronic insomnia for patients with mild to moderate traumatic brain injury (MTBI). MBSR is a standardized protocol of meditation and yoga that has been studied extensively in other populations, however the effects of MBSR have not yet been well studied in the proposed population of service members with a Traumatic Brain Injury (TBI) who are experiencing insomnia.

DETAILED DESCRIPTION:
Randomized, controlled trial with 1:1 randomization (n=50). The control group will receive the usual care for TBI through the clinical program with standard providers based on usual patient evaluation and needs. The intervention group will receive MBSR in addition to the usual care through the TBI program.

The usual care pathway will include physician visits, rehabilitation therapies (PT/OT/ST/et al), and other providers as needed based on recommendations by his or her providers. Some variability will exist, but withholding standard of care would be unethical and standardizing care would be impossible. However, providers will be asked that medications, et al that could affect sleep remain unchanged during the trial period (maximum 12 weeks), which is reasonable given that patients have a chronic injury and no emergent/acute needs based on inclusion/exclusion criteria.

Subjects in a control group will be offered complimentary MBSR after 6 month follow up visit is completed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with mild-to-moderate TBI (as defined by the DoD criteria)
2. Right-handedness
3. Insomnia Severity Index ≥15
4. DEERS eligible at the time of enrollment
5. Not pregnant
6. Male and female subjects 18 to 60 years old
7. Insomnia disorder per DSM-V criteria

Exclusion Criteria:

1. Inability to speak or understand English (because this is a group intervention, it requires a common language)
2. Patients who require assistance with activities of daily living (ADLs)
3. Active practice of meditation and/or yoga or participation in meditation/yoga classes in the last 6 months prior to enrollment
4. Signs or symptoms of upper motor neuron syndrome, any major systemic illness or unstable condition which could interfere with protocol compliance
5. Active psychiatric disease that would interfere with participation in the trial, psychotic features, agitation, or behavioral problems within the last 3 months that could interfere with protocol compliance
6. A history of alcohol/substance abuse or dependence within the past 6 months
7. Any neurosurgical intervention affecting brain parenchyma
8. Unstable seizure activity
9. Concurrent participation in another clinical research trial with investigational drug or previous participation with the last investigational drug administered less than 4 weeks prior to screening
10. Females who are pregnant or planning to become pregnant in 6 months following screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-04-12 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Decrease in total score of Insomnia Severity Index (ISI) scale. | Change in the score at baseline, 2 week follow up post treatment completion, 6 months follow up post treatment completion
  compare change in Insomnia Severity Index (ISI, score range 0-28) scores at baseline, 2 week follow up and 6 month follow up. ISI measures severity of insomnia and calculated by adding the scores for all seven items. Results interpretation: 0-7 = No clinically significant insomnia; 8-14 = Subthreshold insomnia; 15-21 = Clinical insomnia (moderate severity); 22-28 = Clinical insomnia (severe). A 6 point decrease is considered clinically significant improvement in symptoms of insomnia.

SECONDARY OUTCOMES:
Change in cognitive function as measured by NIH toolbox | Change in the score at baseline, 2 week follow up post treatment completion, 6 months follow up post treatment completion
  Compare changes in cognitive assessment measured by National Institute of Health (NIH) Toolbox between the groups and at baseline and 2 week follow up within the group.
Change in PCL-5 (Post Traumatic Stress Disorder Check List-5) score | Change in the score at baseline, 2 week follow up post treatment completion, 6 months follow up post treatment completion
  Compare changes in total scores in PTSD Check List-5 (PCL-5) (range 0-80) scores between the groups at baseline, 2 week follow up and 6 month follow and within the group at time points indicated. PCL-5 measures symptoms of PTSD (post traumatic stress disorder) for initial provisional diagnosis, to monitor symptoms before and after treatment and screening individuals for PTSD so they can be appropriately followed by the clinicians. A total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items. symptom cluster severity scores can be obtained by summing the scores for the items within a given cluster. A provisional PTSD diagnosis can be made by treating each item rated as 2 = "Moderately" or higher as a symptom endorsed, then following the diagnostic rule which requires at least: 1 B item (questions 1-5), 1 C item (questions 6-7), 2 D item
Change in RAND-36 (RAND corporation 36 item Health Survey) score | Change in the score at baseline, 2 week follow up post treatment completion, 6 months follow up post treatment completion
  Compare changes in total scores in RAND corporation 36 item Health Survey (RAND-36 range 0-100 on each item) between the groups at baseline, 2 week follow up and 6 month follow and within the group at time points indicated. RAND-36 measures eight concepts: physical functioning, bodily pain, limitations due to physical health problems, limitations due to emotional or personal problems, emotional well-being, social functioning, energy/fatigue and general health perceptions. It also includes a single item that provides an indication of perceived change in health.Scoring the RAND 36-Item Health Survey is a two-step process. First, precoded numeric values are recoded per the scoring key given in Table 1. Note that all items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved. In
Change in PHQ-9 (Patient Health Questionnaire 9) score | Change in the score at baseline, 2 week follow up post treatment completion, 6 months follow up post treatment completion
  Compare changes in total scores in Patient Health Questionnaire 9 (PHQ-9, score range 0-27) between the groups at baseline, 2 week follow up and 6 month follow and within the group at time points indicated. PHQ-9 assesses depression. Scoring: add up all checked boxes on PHQ-9 For every checked Not at all = 0; Several days = 1;More than half the days = 2; Nearly every day = 3, Interpretation of Total (sum of all items) Score: 1-4 Minimal depression; 5-9 Mild depression; 10-14 Moderate depression; 15-19 Moderately severe depression; 20-27 Severe depression
Change in FSS (Fatigue Severity Scale score) | Change in the score at baseline, 2 week follow up post treatment completion, 6 months follow up post treatment completion
  Compare changes in total scores in Fatigue Severity Scale (FSS, score range 9-63) between the groups at baseline, 2 week follow up and 6 month follow and within the group at time points indicated. The Fatigue Severity Scale (FSS) is a method of evaluating the impact of fatigue on participant. The FSS is a short questionnaire that requires participant to rate their level of fatigue. The FSS questionnaire contains nine statements that rate the severity of participant's fatigue symptoms.A total score of less than 36 suggests that participant may not be suffering from fatigue. A total score of 36 or more suggests that participant may need further evaluation by a physician.
Change in MAAS (Mindful Attention Awareness Scale score) | Change in the score at baseline, 2 week follow up post treatment completion, 6 months follow up post treatment completion
  Compare changes in total scores in Mindful Attention Awareness Scale (MAAS, score range 15-90) between the groups at baseline, 2 week follow up and 6 month follow and within the group at time points indicated. The trait MAAS is a 15-item scale designed to assess a core characteristic of mindfulness, namely, a receptive state of mind in which attention, informed by a sensitive awareness of what is occurring in the present, simply observes what is taking place. This is in contrast to the conceptually driven mode of processing, in which events and experiences are filtered through cognitive appraisals, evaluations, memories, beliefs, and other forms of cognitive manipulation.To score the scale, simply compute a mean (average) of the 15 items. Higher scores reflect higher levels of dispositional mindfulness.
Change in PSS (Perceived Stress Scale) | Change in the score at baseline, 2 week follow up post treatment completion, 6 months follow up post treatment completion
  Compare changes in total scores Perceived Stress Scale (PSS, score range 0-40) between the groups at baseline, 2 week follow up and 6 month follow and within the group at time points indicated. The PSS is a global assessment of an individual's perception of psychological stress during the past month. scores are obtained by reversing the scores on the four positive items, e.g., 0=4, 1=3, 2=2, etc. and then summing across all 10 items. Items 4,5, 7, and 8 are the positively stated items.Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress.
Change in NSI (Neurobehavioral Symptom Inventory scale) score | Change in the score at baseline, 2 week follow up post treatment completion, 6 months follow up post treatment completion
  Compare changes in total scores in Neurobehavioral Symptom Inventory (NSI, range 0-88) between the groups at baseline, 2 week follow up and 6 month follow and within the group at time points indicated. The NSI is widely used in the Department of Defense (DoD) for the evaluation of post-concussive symptoms in service members (SMs). In addition, the Department of Veterans Affairs (VA) uses the NSI in its comprehensive traumatic brain injury (TBI) evaluation. Scores are summed at initial visit and follow up visit. number of symptoms of moderate, severe, and very severe intensity and a list of the specific symptoms in each of these rating categories. Change in individual symptom scores of two or more points in a positive direction consistent with recovery (i.e. very severe to moderate, mild or none; severe to mild or none; moderate to none). Change in individual symptom scores of two or more points indicative of symptom worsening or deterioration.
Any changes in blood biomarkers | Change in the score at baseline, 2 week follow up post treatment completion, 6 months follow up post treatment completion
  Compare any changes in biomarkers - cytokines (il-6, IL-10, TNFa), tau, BDNF, IGF-1, amyloid beta 40/42, and melatonin measured at pg/ml at baseline and 2 week follow up.
Changes in SE- sleep efficiency measured by actigraphy devices and polysomnography. | Change in the score at baseline, 2 week follow up post treatment completion, 6 months follow up post treatment completion
  to compare sleep sleep efficiency in % as calculated by total time asleep/total sleep time determined by actigraphy devices and polysomnography.

CONTACTS AND LOCATIONS:
Locations (1):
- Fort Belvoir Community Hospital, Fort Belvoir, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Johansson B, Bjuhr H, Ronnback L. Mindfulness-based stress reduction (MBSR) improves long-term mental fatigue after stroke or traumatic brain injury. Brain Inj. 2012;26(13-14):1621-8. doi: 10.3109/02699052.2012.700082. Epub 2012 Jul 13. PMID 22794665
- [Background] Azulay J, Smart CM, Mott T, Cicerone KD. A pilot study examining the effect of mindfulness-based stress reduction on symptoms of chronic mild traumatic brain injury/postconcussive syndrome. J Head Trauma Rehabil. 2013 Jul-Aug;28(4):323-31. doi: 10.1097/HTR.0b013e318250ebda. PMID 22688212
- [Background] Hubbling A, Reilly-Spong M, Kreitzer MJ, Gross CR. How mindfulness changed my sleep: focus groups with chronic insomnia patients. BMC Complement Altern Med. 2014 Feb 10;14:50. doi: 10.1186/1472-6882-14-50. PMID 24512477